CLINICAL TRIAL: NCT04037228
Title: Surgical Outcomes of the Accelerometer-based Navigation System for Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: 2017.458
Record Dates: First submitted 2019-06-20; First posted 2019-07-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Arthroplasty; Replacement; Knee; Radiotherapy; Image-Guided

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- KneeAlign 2: Those of the group will be adopt KneeAlign 2: accelerometer-based navigation system at total knee arthroplasty.
  Interventions: Device: KneeAlign 2 system (OrthAlign Inc, Aliso Viejo, California)

INTERVENTIONS:
Device: KneeAlign 2 system (OrthAlign Inc, Aliso Viejo, California) — The KneeAlign 2 system (OrthAlign Inc, Aliso Viejo, California) is an accelerometer-based, portable navigation device for TKA that attempts to combine the alignment accuracy of large-console CAS systems, with the ease of use and convenience of conventional alignment methods. It is used to perform the proximal tibial and distal femoral resections in TKA. It consists of a disposable display console (2 × 4 × 2 inches in size) and a reference sensor, both of which are used for the tibial and femoral resections The display console and reference sensor each contains triaxial accelerometers that communicate wirelessly with one another. Briefly, the tibial jig has 2 primary components (a fixed component and a mobile component) connected by a proximal articulation .The fixed component, with the attached reference sensor, is first pinned to the tibia. The purpose of the fixed component is to account for the movement of the tibia during cutting block alignment.

SUMMARY:
Osteoarthritis (OA) is a very common condition in the elderly population. Treatment for end-stage OA is total knee Replacement (TKR)

DETAILED DESCRIPTION:
Overall the success rate of TKR is very high with high patient satisfaction and outcomes. Survivorship depends on patient selection and surgical techniques. Femoral and tibial component mal-alignment might lead to early failure.

Although recent studies have questioned the significance of overall postoperative mechanical alignment on survivorship, most studies still demonstrate alignment to be a crucial factor in the clinical success of TKA [1]. Ritter et al [2], in a review of 6070 TKAs, noted the risk of aseptic failure to significantly increase with a tibial component orientation less than 90° relatives to the tibial axis and a femoral component orientation greater than 8° of valgus relative to the femoral axis (failure rate, 8.7%).

Berend et al [3], in a review of 3152 TKAs, demonstrated that a tibial varus alignment of greater than 3° increased the odds of implant failure and medial bone collapse by roughly 17 times.

The most commonly used methods of component alignment in TKA are an extramedullary (EM) alignment guide for the tibial resection and an intramedullary (IM) alignment guide for the distal femoral resection. Unfortunately, these "conventional" methods have demonstrated a limited degree of accuracy for both overall mechanical alignment and individual component Method to create an even more accurate resection includes the use computer-assisted navigation technique. In a meta-analysis of 29 studies comparing computer assisted surgical (CAS) to conventional techniques in TKA (Mason et al). The authors found that only 68.2% of TKAs in the conventional group achieved an overall mechanical axis within 3° of neutral (vs 91.0% in the CAS group), 65.9% achieved a femoral varus/valgus alignment within 2° of perpendicular to the femoral mechanical axis (vs 90.4% in the CAS group) and 79.7% achieved a tibial varus/valgus alignment within 2° of perpendicular to the tibial mechanical axis (vs 95.2% in the CAS group).

However, despite these advantages, concerns regarding increased capital costs, operative times, extra pin sites, and the learning curve associated with the use of CAS techniques have continued to limit its widespread acceptance.

Another factor that might have limited its usage is that so far no study has shown the accuracy with CAS can directly lead to a longer survivorship of the implant or a better functional outcome. However, the most surgeon still believes a correct align knee will yield a better function and outcome.

This shed the light to a new navigation device. Iorio et.al [4]The KneeAlign 2 system (OrthAlign Inc, Aliso Viejo, California) is an accelerometer-based, portable navigation device for TKA that attempts to combine the alignment accuracy of large-console CAS systems, with the ease of use and convenience of conventional alignment methods. It is used to perform the proximal tibial and distal femoral resections in TKA. It does not require the use of a large console for registration and alignment feedback and is compatible with any TKA system. It consists of a disposable display console (2 × 4 × 2 inches in size) and a reference sensor, both of which are used for the tibial and femoral resections The KneeAlign 2 is the second version of the KneeAlign originally developed to perform only the proximal tibia resection in TKA. The KneeAlign 2 required the additional design of a femoral jig and cutting block and allows for the use of the same display console to perform both the proximal tibia and distal femur resections. The display console and reference sensor each contains triaxial accelerometers that communicate wirelessly with one another. The surgical technique for using the KneeAlign 2 to perform the tibial resection is the same as previously described Briefly, the tibial jig has 2 primary components (a fixed component and a mobile component) connected by a proximal articulation .The fixed component, with the attached reference sensor, is first pinned to the tibia. The purpose of the fixed component is to account for the movement of the tibia during cutting block alignment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged over 18 years old
* All patients must provide their written consent
* patients with a history of osteoarthritis, rheumatoid arthritis, or post-traumatic arthritis who will receive a primary, posterior-stabilized TKA.
* All patients should have at least 8 years of school education;
* Radiological evidence of osteoarthritis with Kellgren and Lawrence grade 2 or above

Exclusion Criteria:

* Patients are planned to receive a unicondylar or patellofemoral arthroplasty.
* Patients with previous cases of alcoholism or drug abuse;
* Pregnancy and breast-feeding;
* Presence of serious pathologies;
* revision surgery
* Knee infection
* Non-consenting patients who have not provided the written Informed Consent;
* Mechanical instability, ligamentous laxity/deficiency and gross deformity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteoarthritis knee patients in hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Radiological Assessments of the knees at baseline | Through study completion, an average of 1 year
  Standing antero-posterior (AP) hip-knee-ankle (HKA) and lateral knee-to-ankle radiographs will be performed to determine the varus/valgus alignment and the posterior slope of the tibial components relative to the mechanical axis.
Changes of Radiological Assessments of the knees post-operatively | Through study completion, an average of 1 year
  Standing antero-posterior (AP) hip-knee-ankle (HKA) and lateral knee-to-ankle radiographs will be performed to determine the varus/valgus alignment and the posterior slope of the tibial components relative to the mechanical axis.

SECONDARY OUTCOMES:
Knee Functions measure by the Knee Society Score | Through study completion, an average of 1 year
  Questionnaire - Physician will assess on the Visual Analog Scale in pain score (None to Severe), Flexion Contracture (None to >20°), Extension lag (None to 20°), Total Range of Flexion (0-5° to 121-125°), Alignment (0° to Over 15°), Antero-posterior stability (<5mm to 10+mm), Mediolateral stability (<5° to 15°). Patients will record individuals' satisfaction, functional activities, and expectations.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided